CLINICAL TRIAL: NCT01647581
Title: Risk of Post-Polypectomy Bleeding With Prophylactic Hemoclipping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLNB-005-13F; DVAMC-11-026 (Other Grant/Funding Number: MERIT)
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Post-polypectomy Bleeding; Polypectomy; Elective Colonoscopy
Keywords: hemoclip; colonoscopy; post-polypectomy bleed
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clip (Experimental): A clip is been placed at the polypectomy site.
  Interventions: Device: Hemoclip Placement
- No Clip (Placebo Comparator): A hemoclip is not placed at the site of the polypectomy.
  Interventions: Device: NO hemoclip placement

INTERVENTIONS:
Device: Hemoclip Placement — Placement of hemoclip at polypectomy site for polyps at least 1cm in size
  Other Names: Clip
  Arms: Clip
Device: NO hemoclip placement — No hemoclip placement (placebo / sham)
  Other Names: No Clip
  Arms: No Clip

SUMMARY:
A randomized trial aimed at determining whether or not hemoclips are effective in preventing post-polypectomy bleeds on polyps that are 10mm in size or greater.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective colonoscopy

Exclusion Criteria:

* Patients in which polypectomy can not be performed safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11182 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Feagins, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (3):
- United States (3):
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feagins LA, Smith AD, Kim D, Halai A, Duttala S, Chebaa B, Lunsford T, Vizuete J, Mara M, Mascarenhas R, Meghani R, Kundrotas L, Dunbar KB, Cipher DJ, Harford WV, Spechler SJ. Efficacy of Prophylactic Hemoclips in Prevention of Delayed Post-Polypectomy Bleeding in Patients With Large Colonic Polyps. Gastroenterology. 2019 Oct;157(4):967-976.e1. doi: 10.1053/j.gastro.2019.05.003. Epub 2019 May 31. PMID 31158369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11,182 enrolled into the study, but 10,084 screen failures as the majority did not have a polyp 1cm in size to meet criteria for randomization
Pre-assignment Details: Must have polyp 1cm in size removed during colonoscopy
Period: Overall Study
Arm/Group | Clip | No Clip
Started | 547 | 551
Completed | 530 | 520
Not Completed | 17 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clip | No Clip | Total
Number analyzed (Participants) | 530 | 520 | 1050
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 251 | 246 | 497
  >=65 years | 279 | 274 | 553
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.9) | 64.0 (8.6) | 64.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 516 | 499 | 1015
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 370 | 375 | 745
  black | 117 | 110 | 227
  hispanic | 42 | 31 | 73
  other | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 530 | 520 | 1050
smoking [Count of Participants; unit: Participants] | 197 | 190 | 387

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Delayed Post Polypectomy Bleeding
Description: rectal bleeding with associated Hb 2g drop, hemodynamic instability, or need for repeat colonoscopy or angiography or surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clip | No Clip
Number analyzed (Participants) | 530 | 520
Participants | 12 | 15

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Clip | No Clip
All-Cause Mortality (participants affected / at risk) | 1/547 | 1/551
Serious Adverse Events (participants affected / at risk) | 25/547 | 21/551
Other Adverse Events (participants affected / at risk) | 5/547 | 2/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clip (N=547) | No Clip (N=551)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Chest pain / bradycardia (Cardiac disorders) | 3 | 0
Chronic renal failure (Renal and urinary disorders) | 1 | 0
Cerebrovascular accident / Deep vein thrombosis (Vascular disorders) | 2 | 0
Elective laminectomy (Surgical and medical procedures) | 0 | 1
Gallstones (Hepatobiliary disorders) | 0 | 1
Post-polypectomy bleed (Injury, poisoning and procedural complications) | 12 | 15
Post-polypectomy coagulation syndrome (Injury, poisoning and procedural complications) | 0 | 1
Rectal absess (Gastrointestinal disorders) | 1 | 0
Respiratory illnesses and diseases (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Unimportant bleed (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clip (N=547) | No Clip (N=551)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Multiple falls (Injury, poisoning and procedural complications) | 1 | 0
Epistaxis (Blood and lymphatic system disorders) | 0 | 1
Unimportant bleed (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT01647581/Prot_SAP_000.pdf